CLINICAL TRIAL: NCT03668444
Title: Mobile Support to Improve Recovery and Treatment Court Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Live Inspired, LLC (Industry)
Collaborators: The Miriam Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Grant # 1 R41 DA046268-01A1
Record Dates: First submitted 2018-09-11; First posted 2018-09-12 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Substance Use
Keywords: Text Messaging
MeSH Terms: conditions — Substance-Related Disorders | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Who Masked: Outcomes Assessor
Masking Description: Assessors are blinded to conditions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TXS- Supportive Text Group (Experimental): Participants randomized to this arm (TXS) of the study will receive care as usual within the Drug Treatment Court (DTC) system plus supportive daily text messages which will be delivered at specific times each day for 30 days and will be signed by the judge for their specific DTC. (TXS) Group receives text messages for drug treatment compliance.
  Interventions: Behavioral: TXS- Supportive Text Group
- TAU- Treatment As Usual Group (Placebo Comparator): Participants randomized to the (TAU) arm of the study will continue to participate in court-ordered treatments as usual with no additional intervention. Participants will receive motivational text messages for 30-days.
  Interventions: Behavioral: TAU- Treatment As Usual

INTERVENTIONS:
Behavioral: TXS- Supportive Text Group — TXS participants will receive one treatment supportive text message each day for 30 days.These messages will address three domains 1) Recovery oriented messages, 2) Avoiding relapse and sanctions,and 3) Commitment to family, community and the Drug Treatment Court program. After receiving each text message, participants will receive a second message asking them to reply with a rating of how helpful the original message was. Ratings will use a 5-point Likert scale,ranging from 1-not at all helpful to 5-extremely helpful. Participants will also be asked to describe, via text message, what they liked or did not like about the original message, and suggest a better message for those they did not like.
  Other Names: Intervention
  Arms: TXS- Supportive Text Group
Behavioral: TAU- Treatment As Usual — Participants randomized to the TAU arm of the study will continue to participate in court-ordered treatments as usual with no additional intervention. Participants will receive one motivational text message for the 30-days.
  Other Names: Control
  Arms: TAU- Treatment As Usual Group

SUMMARY:
This study will fully develop and implement an interactive text messaging intervention system for individuals sentenced to DTC. Upon completion of programming and testing of messages the investigators will enroll 40 participants and randomize participant to a control condition (TAU Group) or the intervention condition (TXS Group). Assessments will occur at enrollment, and day 30 follow up.

DETAILED DESCRIPTION:
This study builds on pilot work in which Live Inspired LLC and research partners, have a history of collaboration in the development, revision, and evaluation of web-based and mobile phone technologies to promote behavior change. For this project the investigators will fully develop and implement an interactive text messaging intervention system for individuals sentenced to DTC who are entering the program, at which time participants are expected to begin addressing underlying issues related to their addiction, and during which time participants are highly vulnerable to relapse and noncompliance with mandated activities. Outcomes will include participation in and compliance with Court-mandated appointments, abstinence from drug use (measured by urine testing), participation in substance abuse treatment, participation in education/employment training programs, and participation in related programs and workshops as directed by the Court. Data will be collected directly from Court records using a database established by the participating courts for this study.

ELIGIBILITY:
Inclusion Criteria:

To be eligible, participants must be

1. Age >18;
2. Newly enrolled in the drug court program [within 1 month];
3. Own a mobile phone and use text messaging;
4. have a phone plan that allows unlimited texting;
5. Agree to participate in the study protocol and be available for all assessments through the final 30-day assessment; and
6. Speak and read English.

Exclusion criteria:

We will exclude anyone who is not able to participate in the intervention or assessments (e.g., deaf, blind, or otherwise impaired and unable to participate in computerized assessment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility as measured by study completion | 30 day
  Percent of participants completing all assessment.
Acceptability as measured by rating of text messages | 30 days
  Participant ratings of TXS messages for helpfulness and liking.

CONTACTS AND LOCATIONS:
Overall Officials: Ernestine Jennings, PhD, Principal Investigator — The Miriam Hospital

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.